CLINICAL TRIAL: NCT06086184
Title: Pilot Study to Evaluate the Effectiveness of an Acceptance and Commitment Therapy (ACT)-Based Treatment Approach With Inpatient Group Therapy Interventions for Patients With Psychosis Spectrum Disorder
Brief Title: Inpatient Group Acceptance and Commitment Therapy (ACT) for Psychosis Spectrum Disorder
Acronym: ASPIRE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vivantes Netzwerk für Gesundheit GmbH (Other)
Responsible Party: Principal Investigator, Prof. Dr. Andreas Bechdolf, Head of Psychiatry Vivantes Klinikum Am Urban and Klinikum im Friedrichshain, Vivantes Netzwerk für Gesundheit GmbH
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ethik-26/23
Record Dates: First submitted 2023-10-05; First posted 2023-10-17 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Psychotic Disorders; Acceptance and Commitment Therapy; Psychotherapy, Group; Inpatients
Keywords: Mindfulness; Acceptance and Commitment Therapy; Psychotherapy, Group; Inpatients; Psychotic Disorders
MeSH Terms: conditions — Psychotic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ACT group therapy (Experimental): High-frequency inpatient ACT group therapy program for patients with psychosis spectrum disorder.
  Interventions: Behavioral: ACT group therapy

INTERVENTIONS:
Behavioral: ACT group therapy — Participation in four sessions of the inpatient "Compass Group" and eight sessions of the inpatient "Here-and-Now Group". This should be completed within four weeks and may be completed within six weeks in exceptional cases. The groups are designed as a semi-open group with one therapist and one cotherapist each and are integrated into the existing therapy plan.

SUMMARY:
The pilot study that will serve as the basis for the larger project - a multicenter randomized controlled single-blinded trial (RCT) will focus on testing the feasibility and efficacy of an inpatient group ACT treatment program and its effects on symptom severity and patient satisfaction in patients with psychosis spectrum disorder. The ACT-specific treatment program for inpatients with psychosis spectrum disorder is designed to enable patients to deal with their disease in an accepting manner over the long term, to promote self-determined and positive attitudes toward treatment and support options, and thus to reduce rehospitalization rates.

DETAILED DESCRIPTION:
Inpatient hospitalization is an important time to provide patients with psychosis spectrum disorder with skills to better manage symptoms and improve functioning after discharge. The long-term goal is to reduce the negative consequences of these disorders and to have a lasting positive impact on the course of the disease. Against this background, the aim of a larger-scale future study project is to evaluate a specific ACT-based four-week treatment program providing inpatient group therapy interventions for patients with psychosis spectrum disorder. The ACT-specific treatment program is designed to enable patients to deal with their disease in an accepting manner over the long term, to promote self-determined and positive attitudes toward treatment and support options, and thus to reduce rehospitalization rates. The pilot study will focus on testing the feasibility and efficacy of the inpatient group ACT treatment program and its effects on symptom severity and patient satisfaction in patients with psychosis spectrum disorder. Here, treatment will include a high-frequency four-week inpatient ACT group therapy program with a focus on the core ACT process of mindfulness in addition to standard inpatient treatment. Within the scope of the survey, possible side effects of the intervention will also be recorded and mapped by conducting qualitative individual interviews and documenting serious adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Patients with psychosis spectrum disorder with the following diagnoses according to the Diagnostic and Statistical Manual Diploma in Social Medicine 5 ("Schizophrenia Spectrum and Other Psychotic Disorders"):
* Schizophrenia
* Schizophreniform disorder
* Schizoaffective disorder
* Delusional disorder
* Brief psychotic disorder
* Psychotic disorder due to another disorder
* Substance-induced/medication-induced psychotic disorder
* Depressive episode with psychotic symptoms
* Manic or bipolar episode with psychotic symptoms

Exclusion Criteria:

* Patients decline to participate in the treatment program
* Language or intellectual abilities insufficient for study participation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-10-16 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Positive and Negative Syndrome Scale (PANSS) | T0 Baseline Examinations: Before the start of the intervention at study enrollment T1 Final examinations: After the end of the four-week intervention (week 5) T2 Follow-up examinations: 6 months after the end of the intervention
  The primary endpoint symptom severity is assessed using the German version of the established Positive and Negative Syndrome Scale (PANSS). The PANSS consists of a third-party assessment interview in which 30 symptoms are rated using a seven-point scale ranging from 1 (nonexistent) to 7 (extreme symptom). Symptoms are assigned to three scales: The Positive Scale, the Negative Scale, and the General Psychopathology Scale. The PANSS is widely used and is considered the gold standard for assessing psychopathology in people with psychotic disorders because of its good reliability and validity.

SECONDARY OUTCOMES:
Global Assessment of Functioning (GAF) | T0 Baseline Examinations: Before the start of the intervention at study enrollment T1 Final Examinations: After the end of the four-week intervention (week 5) T2 Follow-up Examinations: 6 months after the end of the intervention
  The general level of functioning is assessed using the German version of the Global Assessment of Functioning (GAF) numerical external assessment scale. The GAF is divided into 10 levels of functioning with 10 points each and ranges from 100 (highest level of functioning) to 1 (lowest level of functioning). Environmental conditions and physical illness are explicitly not to be considered here. Mental, social, and occupational functioning are thought of as being on a hypothetical continuum from mental health to illness.
World Health Organization Quality of Life Brief Version (WHOQOL-BREF) | T0 Baseline Examinations: Before the start of the intervention at study enrollment T1 Final Examinations: After the end of the four-week intervention (week 5) T2 Follow-up Examinations: 6 months after the end of the intervention
  Quality of life is measured with the German version of the WHOQOL-BREF (World Health Organization Quality of Life Brief Version), an abbreviated version of the WHOQOL-100 (World Health Organization Quality of Life 100). The WHOQOL-BREF, which is a brief self-report instrument, consists of a total of 26 items, which are assigned to the 4 domains of physical health (7 items), psychological health (6 items), social relationships (3 items) and environmental health (8 items). Two other items measure overall quality of life and general health. Each individual item of the WHOQOL-BREF is scored from 1 to 5 on a response scale, which is stipulated as a five-point ordinal scale (low score of 1 to high score of 5). The average score for each domain is calculated, resulting in an average domain score between 4 and 20. This average domain score is multiplied by 4 to transform it into a scaled score, with a higher score indicating a better quality of life.
Fragebogen für Akzeptanz und Handeln (FAH-II) | T0 Baseline Examinations: Before the start of the intervention at study enrollment T1 Final Examinations: After the end of the four-week intervention (week 5) T2 Follow-up Examinations: 6 months after the end of the intervention
  German version of the Acceptance and Action Questionnaire (AAQ-II). The AAQ-II was developed to measure experience avoidance based on the model of psychological flexibility. It consists of a 7-point Likert scale. Participants rated between 1 (never true) and 7 (always true) how well the statements describe them. The range of scores is between 7 and 49. Higher scores on the scale indicate higher experience avoidance and lower psychological flexibility.
Fragebogen zur Messung der Patientenzufriedenheit (ZUF-8) | T1 Final Examinations: After the end of the four-week intervention (week 5)
  Patient satisfaction at the end of the intervention is assessed using the German version of the self-report scale Client Satisfaction Questionnaire CSQ-8, the ZUF-8 (Questionnaire for the Measurement of Patient Satisfaction). The eight items are formulated as questions and each have four response options, for which 1-4 points are assigned. After reversal of polarity, all eight item values are summed up to the scale value ZUF-8 (theoretical scale range from 8 to 32). High scale values indicate a high level of "satisfaction", low scale values indicate a low level of "satisfaction".
Questionnaire about the Process of Recovery (QPR) | T0 Baseline Examinations: Before the start of the intervention at study enrollment T1 Final Examinations: After the end of the four-week intervention (week 5) T2 Follow-up Examinations: 6 months after the end of the intervention
  The German version of the self-report scale Questionnaire about the Process of Recovery (QPR), the Personal Recovery Questionnaire, serves as an instrument for assessing personal recovery. The QPR comprises 15 items, each of which is rated on a 4-point scale (0 = do not agree at all, 1 = do not agree , 2 = partly agree, 3 = agree, 4 = fully agree ) and has been validated in German.
Comprehensive Inventory of Mindfulness Experiences (CHIME) | T0 Baseline Examinations: Before the start of the intervention at study enrollment T1 Final Examinations: After the end of the four-week intervention (week 5) T2 Follow-up Examinations: 6 months after the end of the intervention
  Mindfulness skills are assessed with the German self-report scale Comprehensive Inventory of Mindfulness Experiences (CHIME). CHIME is a questionnaire for self-assessment of different aspects of mindfulness. It comprises 37 items that are assigned to eight subscales. Items are scored on a 5-point Likert scale ranging from 1 (never) to 5 (very often). The higher the the arithmetic mean the better the mindfulness skills.
Cognitive Fusion Questionnaire (CFQ-D) | T0 Baseline Examinations: Before the start of the intervention at study enrollment T1 Final Examinations: After the end of the four-week intervention (week 5) T2 Follow-up Examinations: 6 months after the end of the intervention
  Cognitive fusion is assessed with the German version of the self-report questionnaire Cognitive Fusion Questionnaire (CFQ). The Cognitive Fusion Questionnaire (CFQ) assesses cognitive fusion, or rigidly following self-generated rules. The CFQ is a 7 item self-report instrument with a range of 7-49. Higher scores are indicative of a higher level of cognitive fusion.

OTHER OUTCOMES:
Number of group therapy sessions attended and drop out rate | Therapy attendance during the four-week intervention will be measured at T1 Final Examinations after the end of the four-week intervention (week 5).
  To provide evidence on the feasibility and acceptability of the intervention, therapy attendance in the ACT-specific group therapy treatment program (reported as number of group therapy sessions attended) and dropouts from study-related treatment (reported as drop out rate in percent) will be recorded.
Qualitative semi-structured interview analysis according to Mayring | T1 Final Examinations: After the end of the four-week intervention (week 5).
  A focused, semi-structured guided interview will be used to explore research questions related to the desirable and undesirable effects of inpatient ACT-specific group therapy.
  The key questions are:
  1. What have ACT group therapies done for you?
  2. Is this effect desired for you?
  3. Did you experience any unwanted effects?
  4. What did you notice about your symptoms during and after ACT group therapy sessions? The qualitative individual interviews are recorded with a recording device and transcribed by the study staff. The evaluation of the transcribed, semi-structured interviews on the desired and undesirable effects of the intervention is carried out using the qualitative content analysis method according to Mayring. The qualitative content analysis according to Mayring is a structured, qualitative method for the systematic and theory-driven evaluation of text-based data.
WHO Alcohol, Smoking and Substance Involvement Screening Test (WHO ASSIST) | T0 Baseline Examinations: Before the start of the intervention at study enrollment T2 Follow-up Examinations: 6 months after the end of the intervention
  Since substance use can have an influence on the development of the measured data to be assessed, substance use will also be systematically recorded.
ACT Fidelity Measure (ACT-FM) | ACT Fidelity Measure will be evaluated during the four-week intervention.
  The raters use a German translation of the ACT Fidelity Measure (ACT-FM), which is validated in English and can be used in different therapy contexts.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Bechdolf, Prof. Dr., Study Director — Senior consultant department of psychiatry Vivantes Klinikum Am Urban and Klinikum im Friedrichshain
Locations (1):
- Vivantes Klinikum Am Urban, Kreuzberg, State of Berlin, Germany